CLINICAL TRIAL: NCT03931577
Title: Effectiveness and Cost-effectiveness of Improving Clinicians' Diagnostic and Communication Skills on Antibiotic Prescribing Appropriateness in Patients With Acute Cough in Primary Care in Catalonia.
Brief Title: Effectiveness of Improving Diagnostic and Communication Skills on Antibiotic Prescribing Appropriateness in Acute Cough
Acronym: ISAAC-CAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Universitat Internacional de Catalunya (Other); Fundacio d'Atencio Primaria (Other); Universitat Pompeu Fabra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P18/227
Record Dates: First submitted 2019-04-08; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Respiratory Tract Infections; Cough
Keywords: Antimicrobial Stewardship; Cost-Benefit Analysis; Anti-Bacterial Agents; Primary Health Care
MeSH Terms: conditions — Respiratory Tract Infections; Cough

STUDY DESIGN:
Intervention Model Description: Cluster randomised factorial controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C-reactive protein rapid testing (Experimental): Continuous (workshop and monthly web-based training) disease-focused intervention with the use of C-reactive protein rapid testing.
  Interventions: Diagnostic Test: C-reactive protein rapid testing
- Enhancement of communication skills (Experimental): Continuous (on-site and monthly online training) illness-focused intervention with enhancement of communication skills to optimise doctor-patient consultations and share decision making with the aid of patient-centred leaflets.
  Interventions: Procedure: Communication skill enhancement
- C-reactive protein + communication skills (Experimental): Continuous (workshop and monthly web-based training) disease-focused intervention with C-reactive protein rapid testing and on-site and continuous (monthly online training illness-focused intervention) with enhancement of communication skills to optimise doctor-patient consultations and share decision making with the aid of patient-centred leaflets.
  Interventions: Diagnostic Test: C-reactive protein rapid testing; Procedure: Communication skill enhancement
- Usual care (No Intervention): Usual care.

INTERVENTIONS:
Diagnostic Test: C-reactive protein rapid testing — Continuous (workshop and monthly web-based training) disease-focused intervention with the provision of CRP rapid testing in the primary care practices.
  Other Names: CRP
  Arms: C-reactive protein + communication skills; C-reactive protein rapid testing
Procedure: Communication skill enhancement — Continuous (on-site and monthly online training) illness-focused intervention (enhancement of communication skills to optimise doctor-patient consultations and share decision making with the aid of patient-centred leaflets) in the primary care practices.
  Other Names: Leaflet provision
  Arms: C-reactive protein + communication skills; Enhancement of communication skills

SUMMARY:
Despite their marginal benefit, about 60% of uncomplicated acute lower respiratory infections (ALRTI) are currently treated with antibiotics. Several strategies have been developed to reduce inappropriate antibiotic prescribing, with the use of point-of-care C-reactive protein (CRP) testing and the improvement of the communication skills being the most effective interventions, but most of the studies have been carried out outside Mediterranean countries. This study is aimed at evaluating the effect of a disease-focused intervention (CRP) and an illness-focused intervention (improvement of communication skills to optimise doctor-patient consultations and share-decision making with the aid of patient-centred leaflets) on antibiotic prescribing for patients with ALRTIs in Catalan primary care by means of a cluster, randomised, factorial, controlled trial. Primary care centres will be assigned to four trial arms: usual care, use of CRP testing, enhanced communication skills backed up with leaflets, or combined interventions. The main outcome will be antibiotic use within the first 6 weeks and the quality adjusted life years. A pharmacoeconomic analysis of the impact of these interventions will be assessed.

DETAILED DESCRIPTION:
Background: Most antibiotics are prescribed in primary care, and most commonly for acute lower respiratory infections (ALRTI). Despite their marginal benefit, about 60% of these infections are currently treated with antibiotics in Catalonia, Spain. Several strategies have been developed to reduce inappropriate antibiotic prescribing, with the use of C-reactive protein (CRP) rapid testing and the improvement of the communication skills being the most effective interventions. However, most studies have been carried out outside Mediterranean countries. This study aims to evaluate the effectiveness and the efficiency of a continuous disease-focused intervention (CRP) and an illness-focused intervention (enhancement of communication skills to optimise doctor-patient consultations and share decision making with the aid of patient-centred leaflets) on antibiotic prescribing in patients with ALRTIs in Catalan primary care centres.

Methods/design: A cluster, randomised, factorial, controlled trial aimed at including 20 primary care centres (n=2,940 patients) with patients older than 18 years presenting for a first consultation with ALRTI, therefore with presence of infected acute cough of up to 3 weeks' duration as the predominant symptom. Centres, according to socioeconomic and antibiotic consumption, will be randomly assigned according to hierarchical clustering to any of four trial arms: usual care, CRP testing, enhanced communication skills backed up with patient leaflets, or combined interventions. A cost-effectiveness and cost-utility analysis will be performed from the perspective of public health system. A qualitative study aimed at identifying the expectations and concerns in patients with ALRTIs and the satisfaction of clinicians with the different interventions will also be performed. Clinicians assigned to the interventions will participate in a 2-hour training workshop before the inception of the trial and will receive a monthly intervention-tailored training module during the trial. Clinical effectiveness will be measured by the antibiotic use within the first 6 weeks and the quality adjusted life years and secondary outcomes will be duration of illness and severity of cough measured with a symptom diary, healthcare reconsultations, hospital admissions and complications. National health care perspective will be adopted and the temporal horizon of the analysis will be one year. Health care costs will be considered and expressed in € of the current year of the analysis. Univariate and multivariate sensitivity analysis will be carried out.

Discussion: The ISAAC-CAT project aims to improve the management of ALRTIs in primary care through use of two different clinicians' skills to help target antibiotic prescribing only to those most likely to benefit, and thereby reduce the risk of unnecessary exposure to antibiotics leading to adverse effects and/or the development of AMR without having a negative impact on health status, thus benefiting individual patients and society at large. This project will contribute to evaluate the effectiveness and efficiency of different strategies for more appropriate antibiotic prescribing that are currently out of the scope of the actual guidelines.

ELIGIBILITY:
Inclusion Criteria:

* age equal or older than 18 years
* first consultation for acute cough (new cough or worsening of a previous cough) as the predominant symptom
* of up to 3 weeks' duration
* which the clinician believes to be an infectious acute lower respiratory tract infection

Exclusion Criteria:

* a working diagnosis of a non-infective disorder, such as heart failure, pulmonary embolus, oesophageal reflux, or allergy
* use of antibiotics in the previous two weeks
* immunological deficiencies, and/or
* inability to provide informed consent or unable to follow the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2940 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Antibiotic use | Day 42
  Number of antibiotics consumed (as documented in the CRFs and double-checked by the Pharmacy Unit of Institut Català de Salut that can track if the antibiotic has been dispensed at any of the Catalan pharmacies)
Health status | Difference between baseline visit and day 42
  Quality of life score obtained using the EuroQol questionnaire

SECONDARY OUTCOMES:
Re-consultations and complications | Day 42
  Number of re-consultation for new or worsening symptoms, new signs, or hospital admission, assessed by review of medical notes (practice staff, the local study team, or both using a standard form to report these data), and Number of complications regarding the ALRTI
Duration of symptoms and duration of severe symptoms | Day 42
  Number of days until symptoms are rated daily as 0 (no problem) (information is reported by patients in self-completed diaries)
Antibiotic prescription at the baseline visit | Baseline visit
  Number of antibiotic prescriptions at the baseline visit, differentiating immediate and delayed antibiotic prescribing, and antibiotic dispensing at the pharmacies
Drugs other than antibiotics | Day 42
  Number of non-antibiotic prescriptions (reported by patients in self-completed diaries)
Tests ordered by clinicians | Day 42
  Number of tests ordered by clinicians (reported in the CRF)
Patient satisfaction with care | Day 14
  Patient satisfaction score reported in the symptom diary. Measured with a question that has used in previous studies: How satisfied are you with the consultation? Range from 0 (nothing satisfied) to 5 (extremely satisfied).
Patient perception of the usefulness of the information received. | Day 14
  Patient perception score about the usefulness of the information received. Measured with a question that has used in previous studies: Do you consider that the information received from your doctor has been useful? Range from 0 (nothing useful) to 5 (extremely useful).
Patient future consulting intention | Day 14
  Patient future consulting intention score. Measured with a question that has used in previous studies: Do you think you will attend the doctor in future occasions in case you present the same symptoms? Range from 0 (totally unlikely) to 5 (sure).
Serious adverse events | Day 42
  Number of serious adverse events (assessed by review of medical notes (practice staff, the local study team, or both using a standard form to report these data)
Absenteeism | Baseline visit
  Number of days of sick leave (collected in the CRFs)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Morros, MD PhD, Study Chair — Clinical pharmacologist
Locations (1):
- La Marina Health Center, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Reposition in SCENTIA
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: First 15 years after publication
Access Criteria: On demand
URL: http://scientiasalut.gencat.cat

REFERENCES:
- [Derived] Medina-Perucha L, Garcia-Sangenis A, Moragas A, Galvez-Hernandez P, Cots JM, Lanau-Roig A, Borras A, Amo I, Monfa R, Llor C, Berenguera A. Autonomy, power dynamics and antibiotic use in primary healthcare: A qualitative study. PLoS One. 2020 Dec 18;15(12):e0244432. doi: 10.1371/journal.pone.0244432. eCollection 2020. PMID 33338078
- [Derived] Ruiz R, Moragas A, Trapero-Bertran M, Siso A, Berenguera A, Oliva G, Borras-Santos A, Garcia-Sangenis A, Puig-Junoy J, Cots JM, Morros R, Mora T, Lanau-Roig A, Monfa R, Troncoso A, Abellana RM, Galvez P, Medina-Perucha L, Bjerrum L, Amo I, Barragan N, Llor C. Effectiveness and cost-effectiveness of Improving clinicians' diagnostic and communication Skills on Antibiotic prescribing Appropriateness in patients with acute Cough in primary care in CATalonia (the ISAAC-CAT study): study protocol for a cluster randomised controlled trial. Trials. 2019 Dec 17;20(1):740. doi: 10.1186/s13063-019-3727-3. PMID 31847912